CLINICAL TRIAL: NCT02440295
Title: Pilot Study to Assess the Use of Spy Elite for Assessment of Amputation Healing
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Principal Investigator, Robert Cuff, Program Director for Integrated Vascular Surgery Residency and Vascular Surgery Fellowship, Corewell Health West
Other Study IDs: 2014-253
Record Dates: First submitted 2015-03-27; First posted 2015-05-12 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Wound Healing; Lower Extremity Amputation; Above Knee Amputation; Below Knee Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower Extremity Amputations: All patients >= 18 years of age requiring Below Knee Amputation (BKA) or Above Knee Amputation (AKA) cared for by the Spectrum Health vascular surgery service will be assessed for eligibility.
  Subjects with a history of allergies to iodides or iodinated contrast agents, pregnant or nursing women, subjects who are unable to provide consent, and prisoners will be excluded. Eighteen subjects will be enrolled in the pilot study. No special population subjects will be enrolled.
  Interventions: Procedure: Lower Extremity Amputation; Device: SPY Elite Imaging System; Drug: Indocyaine Green

INTERVENTIONS:
Procedure: Lower Extremity Amputation
  Other Names: Above Knee Amputation; Below Knee Amputation
Device: SPY Elite Imaging System — The SPY Elite Imaging System is an adjunctive tool that can be used to assess tissue perfusion in real-time and provides surgeons with information that may change their operative plan before leaving the operating room. (http://novadaq.com/products/spy-elite) The system is comprised of two components, the first is the Spy Elite Kit, which is a single-use package containing one 25 mg vial of indocyanine green, one 10 ml vial of sterile Water for injection, and one SPY Elite sterile drape. The second component to the system is the SPY Elite Device which contains a near-infrared light source that illuminates the fluorescent agent within the tissues, an HD video camera captures the intensity of fluorescent marker in real-time, and software that allows the user to capture relative and absolute perfusion values within the surgical field.
  Other Names: SPY Elite Device; SPY Elite Kit
Drug: Indocyaine Green — Indocyaine Green (ICG) is a non-nephrotoxic fluorescent imaging agent with a half-life of 2.5-3 minutes that is administered intravenously.
  Other Names: ICG

SUMMARY:
The purpose of the study is to evaluate the use of the SPY Elite System to assess real-time tissue perfusion of lower extremity amputation sites and to develop parameters to predict healing of amputations at the time of surgery.

This is a pilot study to see if the Spy Elite System is capable of recording accurate measurements on amputation sites to allow some correlation to healing. If this study shows promise for the device, the investigators would plan a larger study in which the data would be assessed in the operating room at time of acquisition and revision performed if needed based on the findings.

DETAILED DESCRIPTION:
The pilot study is a prospective cohort study of consented subjects who require below knee or above knee amputation. The study will start with 18 subjects to assess proof of concept. If a correlation is identified, then a new proposal will be submitted with a larger cohort.

Our hypothesis is that the Spy Elite System can help identify areas of poor tissue perfusion at the time of lower extremity amputation, and predict future potential wound healing complications.

Primary outcome variables include wound healing at 30 days, and intra-operative imaging of amputation sites using the Spy Elite System. Secondary outcome variables include level of amputation, 30-day wound healing complications, readmission rate, need for revision, and subject demographics and co-morbidities.

Subjects who agree to participation will undergo the amputations in the operating suite as per routine. The Spy Elite System will be implemented after final wound closure and prior to dressing placement. A single injection of 10 mg of Indocyanine Green will be administered, followed by 10 ml bolus of normal saline as per manufacturer IFU and recommendations (Attachments B, C, D). Recording from the Spy Elite Device will be saved for analysis. Also, a digital photograph of the surgical wound will be saved for comparison. No changes in operative management based on Spy Elite System will take place in this study.

At subjects routine 30-day follow up appointment, wounds will be assessed for complications, a digital photograph of the incision will be saved, and secondary endpoints will be obtained.

Possible correlations between perfusion values from the Spy Elite System recording and wound healing will be analyzed by the Investigators. The values will not be known until after the photos are taken and the investigators compare ischemic areas to normal areas based on the collected photographs.

ELIGIBILITY:
Inclusion Criteria:

* All patients >= 18 years of age requiring Below Knee Amputation (BKA) or Above Knee Amputation (AKA) cared for by the vascular surgery service will be assessed for eligibility.

Exclusion Criteria:

* Subjects with a history of allergies to iodides or iodinated contrast agents, pregnant or nursing women, subjects who are unable to provide consent, and prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Currently there are no proven, reliable, objective tests to predict wound healing for amputations. Successful wound healing relies heavily on perfusion of the tissue flaps during amputation, which may already be compromised in peripheral vascular patients. Amputation failure results in repeat hospitalizations, surgeries and prolonged immobility for patients. The financial burden for patients and hospitals are significant, as is the psychological and emotional burden for patients facing repeat amputation. Failure rates for BKA and AKA amputations are 10% and 7% respectively. In elderly patients, readmission rates are as high as 27% with a mortality rate of 9% at 30 days.1 With improved ability to identify amputation sites at risk for wound complication and failure, we hope to decrease the need for readmission and repeat surgery.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Wound Healing Post Lower Extremity Amputation | 30 days post
  The primary outcome variable includes wound healing at 30 days and intra-operative imaging of amputation sites using the SPY Elite System.

SECONDARY OUTCOMES:
Level of Amputation | Intra-operative
  The secondary outcome variables include level of amputation.
Wound Healing | 30 days Post Lower Extremity Amputation
  The secondary outcome variables include 30-day wound healing complications.
Readmission Rates | 30 days Post Lower Extremity Amputation
  The secondary outcome variables include readmission rates.
Lower Extremity Amputation Revision | 30 days Post Lower Extremity Amputation
  The secondary outcome variables include need for revision.
Subject Demographics | Participants will be followed for the duration of the hospital stay and 30 days post lower extremity amputation
  The secondary outcome variables include subject demographics
Co-morbidities | Participants will be followed for the duration of the hospital stay and 30 days post lower extremity amputation
  The secondary outcome variables include co-morbidites.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Cuff, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Vogel TR, Petroski GF, Kruse RL. Impact of amputation level and comorbidities on functional status of nursing home residents after lower extremity amputation. J Vasc Surg. 2014 May;59(5):1323-30.e1. doi: 10.1016/j.jvs.2013.11.076. Epub 2014 Jan 7. PMID 24406089
- [Background] Losken A, Zenn MR, Hammel JA, Walsh MW, Carlson GW. Assessment of zonal perfusion using intraoperative angiography during abdominal flap breast reconstruction. Plast Reconstr Surg. 2012 Apr;129(4):618e-624e. doi: 10.1097/PRS.0b013e3182450b16. PMID 22456376
- [Background] Pineda C., Shelton A., Raju N., Welton M. Use of Introperative Fluorescence vascular angiography to assess intestinal perfusion in the creation of intestinal anastomoses. Tech Colo. 2011;15:215-253.
- [Background] Lepow B, Perry D, Armstrong D. The Use of SPY Intra-operative Vascular Angiography as a Predictor of Wound Healing. Podiatry Mgmt. 2011 Aug; 141-148.
- See also: Spy Elite System Overview — http://novadaq.com/products/spy-elite